CLINICAL TRIAL: NCT02159677
Title: Electrical Impedance Myography for the Assessment of Neck and Low Back Pain
Brief Title: Electrical Impedance Myography of Neck and Low Back Pain
Acronym: EIM
Status: Completed | Type: Observational
Sponsor: Skulpt, Inc. (Industry)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: LBP-001-2012; 2R44AR064142 (NIH)
Record Dates: First submitted 2014-06-06; First posted 2014-06-10 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Low Back Pain; Neck Pain
Keywords: EIM
MeSH Terms: conditions — Low Back Pain; Neck Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Healthy Subjects: Healthy subjects aged 21-80 years with no history of present or past disabling back or neck pain, sciatica, cervical radiculopathy, or any generalized neuromuscular condition except for mild polyneuropathy or common mononeuropathies (e.g. carpal tunnel syndrome, ulnar neuropathy at the elbow.) Additionally, subjects cannot have any history of any moderate-to-severe ongoing medical condition producing generalized disability, such as advanced cardiac or renal disease, or metal spine implants of any type.
  Interventions: Device: EIM Measurements
- Radiculopathy Subjects: Subjects aged 21-80 years with a history consistent with radiculopathy based on clinical, radiologic, and standard electrophysiological criteria, as determined by spine expert.
  Interventions: Device: EIM Measurements
- Musculoskeletal Back Pain Subjects: Subjects aged 21-80 years with low back or neck pain without evidence to suggest neuropathic component; i.e. without radiation of pain, sensory loss or weakness.
  Interventions: Device: EIM Measurements
- Undiagnosed Lower Back or Neck Pain Subjects: Subjects aged 21-80 years with a major complaint of lower back or neck pain.
  Interventions: Device: EIM Measurements

INTERVENTIONS:
Device: EIM Measurements

SUMMARY:
The purpose of this study is to assess neck and low back pain using Electrical Impedance Myography (EIM) in order to develop an algorithm to aid primary care providers (PCPs) in the diagnosis of neck/back pain. Secondary goals include the refinement of EIM technology and associated software of ease-of-use and interpretation by PCPs and staff.

ELIGIBILITY:
1. Radiculopathy Subjects:

   Inclusion Criteria:
   * Age 21-80 years old
   * History consistent with radiculopathy based on clinical, radiologic, and standard electrophysiological criteria, as determined by spine expert (Dr. John Keel)

   Exclusion Criteria:
   * Age under 21 or over 80
   * History of a generalized neuromuscular condition, except for mild polyneuropathy or common mononeuropathies (e.g., carpal tunnel syndrome, ulnar neuropathy at the elbow)
   * History of moderate-to-severe ongoing medical conditions producing generalized disability, such as advanced cardiac or renal disease
   * Metal spine implants of any type
2. Musculoskeletal Back Pain Subjects:

   Inclusion Criteria:
   * Age 21 to 80 years old
   * Low back or neck pain without evidence to suggest neuropathic component; i.e., without radiation of pain, sensory loss or weakness

   Exclusion Criteria:
   * Age under 21 or over 80
   * History of sciatica or cervical radiculopathy
   * History of a generalized neuromuscular condition, except for mild polyneuropathy or common mononeuropathies (e.g., carpal tunnel syndrome, ulnar neuropathy at the elbow)
   * History of moderate-to-severe ongoing medical conditions producing generalized disability, such as advanced cardiac or renal disease
   * Metal spine implants of any type
3. Undiagnosed Lower Back or Neck Pain Subjects:

Inclusion Criteria:

* Age 21 to 80 years old
* Major complaint of lower back or neck pain

Exclusion Criteria:

* Age under 21 or over 80
* Recent (<6 month) history of similar symptoms that has been evaluated
* History of a generalized neuromuscular condition, except for mild polyneuropathy or common mononeuropathies (e.g., carpal tunnel syndrome, ulnar neuropathy at the elbow)
* History of moderate-to-severe ongoing medical conditions producing generalized disability, such as advanced cardiac or renal disease
* Metal spine implants of any type

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Neck and Low Back Pain Subjects
Sampling Method: Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Electrical Impedance Myography (EIM) | Screening Visit
  Subjects will undergo EIM testing on the following muscle groups: deltoid, biceps, brachioradialis, triceps, forearm flexors, neck paraspinal muscles, lumbar paraspinal muscles, vastus lateralis, vastus medials, tibialis anterior, extensor hallucis, medial gastrocnemius.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - New England Baptist Hospital, Boston, Massachusetts
  - Skulpt, Inc., Boston, Massachusetts